CLINICAL TRIAL: NCT00095589
Title: Detection of Bladder Cancer by Microsatellite Analysis (MSA) of Urinary Sediment: Multi-Institutional Study
Brief Title: Microsatellite Analysis of Urinary Sediment in Detecting Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0382; U01CA084968 (NIH); P30CA006973 (NIH); 03-12-30-05 (Other: JHM IRB); CDR0000401496 (Other: other); NCT00185627 (obsolete NCT alias)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Microarray Analysis; Cystoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: loss of heterozygosity analysis
Genetic: microarray analysis
Genetic: microsatellite instability analysis
Other: cytology specimen collection procedure
Other: laboratory biomarker analysis
Procedure: computed tomography
Procedure: cystoscopy

SUMMARY:
RATIONALE: New diagnostic procedures such as microsatellite analysis of sediment in the urine may improve the ability to detect bladder cancer without invasive procedures.

PURPOSE: Diagnostic trial to study the effectiveness of microsatellite analysis of sediment in the urine in detecting bladder cancer in healthy participants, participants who have genitourinary conditions requiring cystoscopy, and patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the sensitivity and specificity of microsatellite analysis (MSA) of urine sediment with cystoscopy and urine cytology for detecting bladder cancer in participants undergoing cystoscopy.

Secondary

* Determine the temporal performance characteristics of MSA in urine sediment from these participants.
* Determine which of the 15 individual markers or combination of markers that make up the MSA test are most predictive of the presence of bladder cancer in these participants.

OUTLINE: This is a single-blind, multicenter, cohort study.

Urine and blood specimens are collected from all participants at baseline. Urine specimens are examined using microsatellite analysis, urine cytology, and urinalysis. Patients in groups 2 and 3 also undergo cystoscopy at baseline.

Patients in group 3 undergo cystoscopy, upper tract imaging (e.g., abdominal CT scan), microsatellite analysis, urine cytology, and urinalysis every 3 months for 2 years in the absence of progressive disease.

Microsatellite analysis, which identifies loss of heterozygosity using polymerase chain reaction technique, is conducted for 15 markers: D4S243, D21S1245, FGA, D17S695, D16S476, D9S171, IFN-A, D20S48, D13S802, D17S654, D16S310, THO1, D9S162, D9S747, and MBP.

PROJECTED ACCRUAL: A total of 500 participants (100 each for groups 1 and 2 and 300 for group 3) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Group 1 (healthy volunteers):

  * No prior or concurrent urologic disease or devices
  * No genitourinary (GU) complaints, including urgency or frequency of urination
  * Normal urinalysis and urine cytology
  * Never smoked cigarettes regularly (i.e., ≥ 1 cigarette/day for ≥ 1 year)
  * No suspected exposure to environmental bladder carcinogens for > 1 year, including, but not limited to, the following occupations or exposures:

    * Aluminum industry
    * Aromatic amines
    * Coal gasification
    * Coal tars and pitches
    * Coke plant
    * Dye industry
    * Leather industry
    * Machinist
    * Painter
    * Rubber industry
    * Truck, bus, or taxi drivers
* Group 2 (participants with condition(s) that lead to false-positive urinary bladder cancer screening studies):

  * GU complaints requiring cystoscopy
  * No current GU malignancy
  * At least 1 of the following conditions:

    * Benign prostatic hypertrophy (International Prostate Symptom Score > 12)
    * Foreign bodies (stones, stents, or catheters)
    * Hematuria (gross or microscopic)
    * GU infection (e.g., prostatitis, urinary tract infection, pyelonephritis, urethritis) within the past 3 months and completed treatment

      * No sign of infection at the time of study participation
* Group 3 (superficial bladder cancer patients):

  * Histologically confirmed superficial bladder urothelial malignancy

    * Primary or recurrent disease
  * No nontransitional cell carcinoma of the bladder, upper tract tumors, muscle-invasive tumors, or superficial disease for which local therapy is not appropriate

PATIENT CHARACTERISTICS:

Age

* Over 40

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* See Disease Characteristics

Other

* No prior cancer except nonmelanoma dermatologic malignancy

  * Prior bladder cancer allowed for group 3 patients

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

  * Prior intravesical therapy for bladder cancer allowed for group 3 patients

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. Schoenberg, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (13):
- United States (12):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Stanford Cancer Center, Stanford, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Grand Strand Urology, LLP, Myrtle Beach, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario, Canada